CLINICAL TRIAL: NCT03056534
Title: Post-Approval Study of the R3 Biolox Delta Ceramic Acetabular System - US
Brief Title: R3 Delta Ceramic Acetabular System PAS U.S.
Acronym: R3-PAS
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-4565-10
Record Dates: First submitted 2017-02-06; First posted 2017-02-17 (Actual); Results first posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2024-02

CONDITIONS: Degenerative Joint Disease
Keywords: Primary Total Hip Arthroplasty; Non-Inflammatory Arthritis; Degenerative Joint Disease; R3 Delta Ceramic Acetabular Insert
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: R3 Biolox Delta Ceramic Acetabular System — All study related procedures with the R3 delta Ceramic Acetabular System must be performed according to the recommended surgical technique described in the labeling and in the instructions for use (IFU).

SUMMARY:
R3 Delta Post-Approval Study U.S.

DETAILED DESCRIPTION:
Post-Approval Study of the R3 Biolox Delta Ceramic Acetabular System - US The R3 Ceramic Acetabular System is indicated for use in skeletally mature patients requiring primary total hip arthroplasty due to non-inflammatory arthritis (degenerative joint disease) such as osteoarthritis, avascular necrosis, or traumatic arthritis. The expected timeline for the study is a total of approximately 5 years: 6 months for site initiation, 12 months for subject enrollment, 3 years until the last subject enrolled has reached the 3 year follow-up interval.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18-75 years old and he/she is skeletally mature
* Patient requires primary total hip arthroplasty due to non-inflammatory degenerative joint disease (degenerative joint disease) such as osteoarthritis, avascular necrosis, or traumatic arthritis.
* Patient has met an acceptable preoperative medical clearance and is free from or treated for cardiac, pulmonary, hematological, etc., conditions that would pose excessive operative risk
* Patient is willing and able to participate in required follow-up visits and to complete study procedures and questionnaires
* Patient has consented to participating in the study by signing the IRB/EC approved informed consent form

Exclusion Criteria:

* Patients with insufficient quantity or quality of bone support; metabolic bone disease; osteoporosis
* Patients with neurological or muscular conditions that would place extreme load or instability upon the hip joint
* Patients with active joint infections or chronic systemic infection
* Obese patients where obesity is defined as BMI ≥ 40
* Skeletal immaturity
* Known allergy to implant materials

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: To eliminate the potential for selection bias, Investigators should consecutively pre-screen all subjects undergoing planned total hip replacement with the R3 delta Ceramic Acetabular System.
Sampling Method: Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Foundation for Orthopaedic Research and Education, Tampa, Florida
  - Emory University, Tucker, Georgia
  - Luminis Health, Annapolis, Maryland
  - Rubin Institute for Advanced Orthopedics, Sinai Hospital, Baltimore, Maryland
  - Reno Orthopaedic Clinic Foundation, Reno, Nevada
  - University of Pennsylvania, Department of Orthopaedic Surgery, Philadelphia, Pennsylvania
  - St. David's Center for Hip and Knee Replacement, Austin, Texas
  - INOV8 Healthcare, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 232 participants were screened with 189 participants enrolled to the study at 10 sites; however, 3 sites were terminated early due to lack of enrollment.
Groups:
- R3™ Biolox® Delta Ceramic Acetabular System: Participants that underwent primary total hip arthroplasty with the R3™ Biolox® delta Ceramic Acetabular System
Period: Overall Study
Arm/Group | R3™ Biolox® Delta Ceramic Acetabular System
Started | 189
Completed | 131
Not Completed | 58
Not completed — Participant withdrew consent | 8
Not completed — Participant not able to return | 6
Not completed — Lost to Follow-up | 37
Not completed — Investigator judgment | 1
Not completed — Death | 4
Not completed — Adverse Event | 1
Not completed — Screen fail due to femoral stem implanted not being allowed per protocol | 1

BASELINE CHARACTERISTICS:
Arm/Group | R3™ Biolox® Delta Ceramic Acetabular System
Number analyzed (Participants) | 189
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.60 (12.75)
Age, Customized [Count of Participants; unit: Participants]
  Age Group: < 65 | 112
  Age Group: >= 65 | 77
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110
  Male | 79
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 3
  Race: Black | 37
  Race: White | 146
  Race: Other | 3
Region of Enrollment [Number; unit: participants]
  United States | 189
Operative Side [Count of Participants; unit: Participants]
  Left | 88
  Right | 101
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.00 (5.01)

OUTCOME MEASURES:

1. Primary Outcome: Overall Study Success at 3 Years Postoperative
Description: Number of participants with overall study success were identified as "Success" or "Failure" where success indicated all the following:
  * No component revision for any reason
  * Modified Harris Hip Score (mHHS) greater than or equal to 80 points
  * No radiographic failure (Radiographic failure was defined as no radiolucencies greater than 2 millimeters (mm) in 50% or more in any of the cup or stem zones, no femoral or acetabular subsidence greater than or equal to 5 mm from baseline, and no acetabular cup inclination changes greater than 4 degrees from baseline when accompanied by a "Mild", "Moderate", "Marked" or "Disabled" mHHS pain score.)
Time Frame: 3 Years Postoperative
Population: Overall number of participants with data collected for the time frame indicated.
Measure: Count of Participants; unit: Participants
Arm/Group | R3™ Biolox® Delta Ceramic Acetabular System
Number analyzed (Participants) | 113
Participants
  Success | 100
  Failure | 13

2. Primary Outcome: Component Revisions at 3 Years Postoperative
Description: Number of participants component revisions identified as "Success" or "Failure" with success defined as no component revision for any reason.
Time Frame: 3 Years Postoperative
Population: Overall number of participants with data collected for the time frame indicated.
Measure: Count of Participants; unit: Participants
Arm/Group | R3™ Biolox® Delta Ceramic Acetabular System
Number analyzed (Participants) | 136
Participants
  Success | 135
  Failure | 1

3. Primary Outcome: Number of Participants With Modified Harris Hip Score Greater Than or Equal to 80 Points
Description: The Harris Hip Score (HHS) is a joint specific score that consists of 10 items covering domains of pain, function, functional activities, absence of deformity, and hip range of motion. The modified Harris Hip Score (mHHS) includes all the same domains as the HHS except for the hip range of motion. Total mHHS scale ranges from 0 (worst) to 95 (best). The number of participants were identified as "Success" or "Failure" with success defined as a mHHS that is greater than or equal to 80 points.
Time Frame: 3 Years postoperative
Population: Overall number of participants with data collected for the time frame indicated.
Measure: Count of Participants; unit: Participants
Arm/Group | R3™ Biolox® Delta Ceramic Acetabular System
Number analyzed (Participants) | 124
Participants
  Success | 114
  Failure | 10

4. Primary Outcome: Overall Radiographic Success at 3 Years Postoperative
Description: Number of participants with overall radiographic success identified as "Success" or "Failure" where success indicated all of the following:
  * No radiolucencies greater than 2 millimeters (mm) in 50% or more in any of the cup or stem zones
  * No femoral or acetabular subsidence greater than or equal to 5 mm from baseline
  * No acetabular cup inclination changes greater than 4 degrees from baseline when accompanied by a "Mild", "Moderate", "Marked" or "Disabled" mHHS pain score
Time Frame: 3 Years Postoperative
Population: Overall number of participants with data collected for the time frame indicated.
Measure: Count of Participants; unit: Participants
Arm/Group | R3™ Biolox® Delta Ceramic Acetabular System
Number analyzed (Participants) | 108
Participants
  Success | 106
  Failure | 2

5. Primary Outcome: Number of Participants With Absence of Radiolucency at 3 Years Postoperative
Description: Number of participants identified as "Success" or "Failure" with success defined as no radiolucencies greater than 2 millimeters (mm) in 50% or more in any of the cup or stem zones
Time Frame: 3 Years postoperative
Population: Overall number of participants with data collected for the time frame indicated.
Measure: Count of Participants; unit: Participants
Arm/Group | R3™ Biolox® Delta Ceramic Acetabular System
Number analyzed (Participants) | 119
Participants
  Success | 119
  Failure | 0

6. Primary Outcome: Number of Participants With Absence of Femoral Subsidence or Acetabular Migration at 3 Years Postoperative
Description: Number of participants identified as "Success" or "Failure" with success defined as no femoral subsidence or acetabular migration greater than or equal to 5 millimeters (mm) from baseline.
Time Frame: 3 Years postoperative
Population: Overall number of participants with data collected for the time frame indicated.
Measure: Count of Participants; unit: Participants
Arm/Group | R3™ Biolox® Delta Ceramic Acetabular System
Number analyzed (Participants) | 119
Participants
  Success | 119
  Failure | 0

7. Primary Outcome: Number of Participants With Absence of Acetabular Cup Inclination Changes Greater Than 4 Degrees From Baseline at 3 Years Postoperative
Description: Number of participants identified as "Success" or "Failure" with success defined as no acetabular cup inclination changes greater than 4 degrees from baseline when accompanied by a "Mild", "Moderate", "Marked" or "Disabled" mHHS pain score.
Time Frame: 3 Years postoperative
Population: Overall number of participants with data collected for the time frame indicated.
Measure: Count of Participants; unit: Participants
Arm/Group | R3™ Biolox® Delta Ceramic Acetabular System
Number analyzed (Participants) | 108
Participants
  Success | 106
  Failure | 2

8. Secondary Outcome: Modified Hip Harris Score (mHHS)
Description: The Harris Hip Score (HHS) is a joint specific score that consists of 10 items covering domains of pain, function, functional activities, absence of deformity, and hip range of motion. The modified Harris Hip Score (mHHS) includes all the same domains as the HHS except for the hip range of motion. Total mHHS scale ranges from 0 (worst) to 95 (best).
Time Frame: Preoperative, 3 months, 1 year, 2 years, 3 years
Population: Overall number of participants with data collected for the time frame indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | R3™ Biolox® Delta Ceramic Acetabular System
Number analyzed (Participants) | 184
score on a scale
  Preoperative | 47.60 (11.52)
  3 months: number analyzed (Participants) | 162
  3 months | 89.60 (10.93)
  1 year: number analyzed (Participants) | 145
  1 year | 91.10 (12.02)
  2 years: number analyzed (Participants) | 137
  2 years | 93.00 (10.37)
  3 years: number analyzed (Participants) | 124
  3 years | 93.50 (8.97)

9. Secondary Outcome: Radiographic Findings: Number of Participants With Absence of Radiolucency
Description: The number of participants identified as either "Success" or "Failure" with success defined as no radiolucencies greater than 2 millimeters (mm) in 50% or more in any of the cup or stem zones when accompanied by a "Mild", "Moderate", "Marked" or "Disabled" pain modified Harris Hip Score (mHHS).
Time Frame: 3 months, 1 year, 2 years
Population: Overall number of participants with data collected for the time frame indicated.
Measure: Count of Participants; unit: Participants
Arm/Group | R3™ Biolox® Delta Ceramic Acetabular System
Number analyzed (Participants) | 156
Participants
  3 months: Success | 155
  3 months: Failure | 1
  1 year: number analyzed (Participants) | 142
  1 year: Success | 142
  1 year: Failure | 0
  2 years: number analyzed (Participants) | 135
  2 years: Success | 135
  2 years: Failure | 0

10. Secondary Outcome: Radiographic Findings: Number of Participants With Absence of Femoral Subsidence or Acetabular Migration
Description: The number of participants identified as either "Success" or "Failure" with success defined as no femoral subsidence or acetabular migration greater than or equal to 5 millimeters (mm) from baseline when accompanied by a "Mild", "Moderate", "Marked" or "Disabled" pain modified Harris Hip Score (mHHS).
Time Frame: 3 months, 1 year, 2 years
Population: Overall number of participants with data collected for the time frame indicated.
Measure: Count of Participants; unit: Participants
Arm/Group | R3™ Biolox® Delta Ceramic Acetabular System
Number analyzed (Participants) | 156
Participants
  3 months: Success | 156
  3 months: Failure | 0
  1 year: number analyzed (Participants) | 142
  1 year: Success | 142
  1 year: Failure | 0
  2 years: number analyzed (Participants) | 135
  2 years: Success | 135
  2 years: Failure | 0

11. Secondary Outcome: Radiographic Findings: Number of Participants With Absence of Acetabular Cup Inclination Changes
Description: Number of participants identified as "Success" or "Failure" with success defined as no acetabular cup inclination changes greater than 4 degrees from baseline when accompanied by a "Mild", "Moderate", "Marked" or "Disabled" pain modified Harris Hip Score (mHHS).
Time Frame: 3 months, 1 year, and 2 years
Population: Overall number of participants with data collected for the time frame indicated.
Measure: Count of Participants; unit: Participants
Arm/Group | R3™ Biolox® Delta Ceramic Acetabular System
Number analyzed (Participants) | 141
Participants
  3 months: Success | 137
  3 months: Failure | 4
  1 year: number analyzed (Participants) | 130
  1 year: Success | 127
  1 year: Failure | 3
  2 years: number analyzed (Participants) | 125
  2 years: Success | 122
  2 years: Failure | 3

12. Secondary Outcome: Implant Survivorship Kaplan-Meier Estimate
Description: The Kaplan-Meier estimate of implant survivorship was measured from date of surgery to date of final visit with survival defined as no revision for any reason. A revision indicated reoperation was needed where any component (acetabular cup, acetabular liner, femoral head, or femoral stem) was replaced.
Time Frame: Postoperatively, up to 3 years
Population: Overall number of participants with data collected for the time frame indicated.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | R3™ Biolox® Delta Ceramic Acetabular System
Number analyzed (Participants) | 187
percentage of participants | 99.4 [96.1 to 99.9]

ADVERSE EVENTS:
Time Frame: Adverse events were collected upon implantation of device through study completion, up to 3 years.
Arm/Group | R3™ Biolox® Delta Ceramic Acetabular System
All-Cause Mortality (participants affected / at risk) | 4/189
Serious Adverse Events (participants affected / at risk) | 70/189
Other Adverse Events (participants affected / at risk) | 101/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | R3™ Biolox® Delta Ceramic Acetabular System (N=189)
Left Knee Osteoarthristis (Musculoskeletal and connective tissue disorders) | 2 — Unrelated to device
INTRAOPERATIVE PERIPROSTHETIC FRACTURE OF RIGHT FEMUR (Injury, poisoning and procedural complications) | 1 — SADE, Procedure related
FALL AND DELIRIUM DUE TO HYPONATREMIA (Nervous system disorders) | 1 — Unrelated to device
INCREASED SHORTNESS OF BREATH, HYPOTENSION (Vascular disorders) | 1 — Unrelated to device
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 — Unrelated to device
RIGHT BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Unrelated to device
ANAPHYLACTIC REACTION TO LEFT KNEE INJECTION (Vascular disorders) | 1 — Unrelated to device
DENTAL PAIN (General disorders) | 1 — Unrelated to device
RIGHT KNEE ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
RIGHT HIP ARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 — Unrelated to device
INGUINAL HERNIA (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
ILEITIS (Gastrointestinal disorders) | 1 — Unrelated to device
SEVERE DEGENERATIVE JOINT DISEASE, LEFT HIP (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
OSTEOARTHRITIS LEFT HIP (Musculoskeletal and connective tissue disorders) | 2 — Unrelated to device
PAIN IN RIGHT WRIST (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
CELLULITIS OF RIGHT LOWER LEG (Injury, poisoning and procedural complications) | 1 — Unrelated to device
RECURRENT DISLOCATION OF LEFT TOTAL HIP ARTHROPLASTY (Musculoskeletal and connective tissue disorders) | 1 — SADE, Procedure related
BILATERAL EYE CATARACT (Eye disorders) | 1 — Unrelated to device
OSTEOARTHRITIS LEFT KNEE (Musculoskeletal and connective tissue disorders) | 2 — Unrelated to device
LEFT EYE PAIN, CORNEAL EROSION (Eye disorders) | 1 — Unrelated to device
CALCULUS OF GALLBLADDER WITH ACUTE CHOLECYSTITIS (Blood and lymphatic system disorders) | 1 — Unrelated to device
LEFT-SIDED NUMBNESS AND WEAKNESS (Injury, poisoning and procedural complications) | 1 — Unrelated to device
LEFT HIP OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 4 — Unrelated to device
RIGHT SHOULDER ROTATOR CUFF ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
SEIZURE, ENCEPHALOPATHY (Nervous system disorders) | 2 — Unrelated to device
LEFT AND RIGHT KNEE PAIN (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
CLOSED FRACTURE OF DISTAL END OF RIGHT FIBULA (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
SEVERE DEGENERATIVE JOINT DISEASE, RIGHT HIP (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
MELANOMA, NOSE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Unrelated to device
CARDIOMYOPATHY (Cardiac disorders) | 1 — Unrelated to device
HYPERTROPHIC OBSTRUCTIVE CARDIOMYOPATHY, ATRIAL FIBRILLATION (Cardiac disorders) | 1 — Unrelated to device
LEAD NOISE ON RV (Cardiac disorders) | 1 — Unrelated to device
CHEST WALL HEMATOMA AT PACEMAKER SITE (Injury, poisoning and procedural complications) | 1 — Unrelated to device
LOW BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 — Unrelated to device
LEFT SHOULDER IMPINGEMENT, ACROMIOCLAVICULAR JOINT ARTHROSIS, BICEPS TENDINITIS AND ROTATOR CUFF FRA (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
RIGHT SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
SYPHILIS (Reproductive system and breast disorders) | 1 — Unrelated to device
DEGENERATIVE ARTHRITIS, RIGHT KNEE (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
ATRIAL FLUTTER (Cardiac disorders) | 1 — Unrelated to device
LUMBAR STENOSIS (Nervous system disorders) | 1 — Unrelated to device
OSTEOARTHRITIS, RIGHT HIP (Musculoskeletal and connective tissue disorders) | 2 — Unrelated to device
ACUTE CHOLECYSTITIS (Gastrointestinal disorders) | 1 — Unrelated to device
RIGHT HIP PAIN AND DISCOMFORT (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
SOLITARY BRAIN METASTASIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Unrelated to device
LUNG CANCER, LEFT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Unrelated to device
CHEST PAIN (General disorders) | 1 — Unrelated to device
BILATERAL PTOSIS OF UPPER EYELIDS (Eye disorders) | 1 — Unrelated to device
RIGHT HIP DISLOCATION, CONTUSION OF RIGHT THUMB WI (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
LEFT HIP POSTOPERATIVE PAIN (Injury, poisoning and procedural complications) | 1 — Unrelated to device
UPPER GASTROINTESTINAL BLEEDING (Gastrointestinal disorders) | 1 — Unrelated to device
LEFT HIP ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
GANGLION CYST OF TENDON SHEATH OF RIGHT HAND (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
LEFT HIP PAIN SECONDARY TO OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 — Unrelated to device
FAILED TOTAL HIP JOINT (RIGHT SIDE) (Product Issues) | 1 — Unrelated to device
PERICOLONIC ABSCESS S/P APPENDECTOMY (Gastrointestinal disorders) | 1 — Unrelated to device
ACUTE NONPERFORATED APPENDICITIS (Gastrointestinal disorders) | 1 — Unrelated to device
SPINAL STENOSIS (Nervous system disorders) | 1 — Unrelated to device
OSTEOARTHRITIS, LEFT KNEE (Musculoskeletal and connective tissue disorders) | 2 — Unrelated to device
PATIENT DIAGNOSED WITH CANCER, AGGRESSIVE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Unrelated to device
PRIMARY OSTEOARTHRITIS LEFT HIP (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Unrelated to device
CALCAR FRATURE INTRAOPERATIVELY (Injury, poisoning and procedural complications) | 1 — SADE, Procedure related
LEFT HIP OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 — Unrelated to device
GLENOHUMERAL JOINT OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
LEFT HIP OSTEOARTHRITIS - WORSENING PAIN (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 — Unrelated to device
KNEE OSTEOARTHRITIS, BILATERAL (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
TYPHOID FEVER - PNEUMONIA (Infections and infestations) | 1 — Unrelated to device
SEVERE RIGHT HIP OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 — Unrelated to device
HIP OSTEOARTHRITIS (LEFT HIP) (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
LEFT KNEE OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 — Unrelated to device
BRAIN TUMOR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Unrelated to device
RIGHT HIP ARTHROPLASTY (TOTAL) FOR AVN (AVASCULAR (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
AVASCULAR NECROSIS OF BONE OF LEFT HIP (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
GASTRITIS WITH NAUSEA AND VOMITING (Gastrointestinal disorders) | 1 — Unrelated to device
RIGHT TOTAL KNEE REPLACEMENT (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
DEATH DUE TO DRUG OVERDOSE (Injury, poisoning and procedural complications) | 1 — Unrelated to device
RIGHT INTRAOPERATIVE CALCAR FRACTURE (Musculoskeletal and connective tissue disorders) | 1 — SADE, Procedure related
LEFT TOTAL KNEE REPLACEMENT DUE TO POST-TRAUMATIC (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
OSTEOARTHRITIS IN RIGHT HIP (Musculoskeletal and connective tissue disorders) | 2 — Unrelated to device
SWELLING LEFT IN HIP (Musculoskeletal and connective tissue disorders) | 1 — SADE, Procedure related
BILIARY COLIC (Gastrointestinal disorders) | 1 — Unrelated to device
BILATERAL SHOULDER ARTHRITIS (Nervous system disorders) | 1 — Unrelated to device
CERVICAL MYELORADICULOPATHY (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
END STAGE RIGHT SHOULDER ARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 — Unrelated to device
PELVIC AND LEFT HUMERUS FRACTURES DUE TO FALL (Injury, poisoning and procedural complications) | 1 — Unrelated to device
WORSENING LEFT KNEE OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
WORSENING LEFT HIP OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
WORSENING RIGHT HIP OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
BILATERAL HIP PAIN DUE TO ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 — Unrelated to device
HERNIA (Gastrointestinal disorders) | 1 — Unrelated to device
WORSENING NEPHROTIC SYNDROME (Renal and urinary disorders) | 1 — Unrelated to device
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | R3™ Biolox® Delta Ceramic Acetabular System (N=189)
L KNEE OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
INTRAOPERATIVE PERIPROSTHETIC FRACTURE OF RIGHT FEMUR (Injury, poisoning and procedural complications) | 1
PAIN RIGHT HIP (Injury, poisoning and procedural complications) | 1
FALL AND DELIRIUM DUE TO HYPONATREMIA. (Nervous system disorders) | 1
INCREASED SHORTNESS OF BREATH, HYPOTENSION (Vascular disorders) | 1
SUPERFICIAL PROXIMAL WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1
IT BAND TIGHTNESS (LEFT) (Musculoskeletal and connective tissue disorders) | 1
RADICULAR PAIN, LEFT HIP/LEG (Nervous system disorders) | 1
OCCASIONAL ACHE AT TIP OF STEM (Injury, poisoning and procedural complications) | 1
PAIN, LEFT HIP (Musculoskeletal and connective tissue disorders) | 1
ANAPHYLACTIC REACTION TO LEFT KNEE INJECTION (Vascular disorders) | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1
RAISED PROSTATE SPECIFIC ANTIGEN (Vascular disorders) | 1
RECURRENT DISLOCATION OF LEFT TOTAL HIP ARTHROPLASTY (Musculoskeletal and connective tissue disorders) | 1
RHEUMATOID FLARES (Musculoskeletal and connective tissue disorders) | 1
RIGHT ANKLE PAIN (Musculoskeletal and connective tissue disorders) | 1
SYNCOPE (Cardiac disorders) | 1
HYPERLIPIDEMIA (Metabolism and nutrition disorders) | 2
LEAD NOISE ON RV (Cardiac disorders) | 1
MILD DISCOMFORT RIGHT HIP TROCHANTER REGION (Injury, poisoning and procedural complications) | 1
LEFT HIP ARTHRITIS (Musculoskeletal and connective tissue disorders) | 2
CHEST WALL HEMATOMA AT PACEMAKER SITE (Injury, poisoning and procedural complications) | 1
RIGHT ANKLE SPRAIN, RIGHT GASTROCNEMIUS STRAIN (Injury, poisoning and procedural complications) | 1
RIGHT BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LEFT KNEE ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
CARDIOMYOPATHY (Cardiac disorders) | 1
HYPERTROPHIC OBSTRUCTIVE CARDIOMYOPATHY, ATRIAL FIBRILLATION (Cardiac disorders) | 1
URINARY TRACT INFECTION (Infections and infestations) | 3
ATRIAL FLUTTER (Cardiac disorders) | 1
HYPERTENSION (Vascular disorders) | 1
HYPERCHOLESTEROLEMIA (Metabolism and nutrition disorders) | 1
SEVERE DEGENERATIVE JOINT DISEASE, LEFT HIP (Musculoskeletal and connective tissue disorders) | 1
FULL BODY HIVES (Skin and subcutaneous tissue disorders) | 1
ACUTE NON-RECURRENT SINUSITIS (Infections and infestations) | 1
ANEMIA (Blood and lymphatic system disorders) | 1
ELEVATED LOW DENSITY LIPOPROTEIN LEVEL (Metabolism and nutrition disorders) | 1
ACUTE SINUSITIS (Infections and infestations) | 1
CARDIAC ARRYTHMIAS (Cardiac disorders) | 2
IRON DEFICIENCY ANEMIA (Blood and lymphatic system disorders) | 1
OSTEOARTHRITIS LEFT HIP (Musculoskeletal and connective tissue disorders) | 2
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1
SQUEAKING, LEFT HIP (Injury, poisoning and procedural complications) | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 1
LUMBAR RADICULOPATHY (Nervous system disorders) | 3
ACUTE LEFT HIP PAIN, LUMBAR STRAIN (Injury, poisoning and procedural complications) | 1
LEFT HIP PSOAS TENDINITIS (Musculoskeletal and connective tissue disorders) | 1
BLUNT CHEST TRAUMA, SUBACUTE RIB FRACTURES (Injury, poisoning and procedural complications) | 1
CELLULITIS OF RIGHT LOWER LEG (Injury, poisoning and procedural complications) | 1
BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 1
ACUTE PANSINUSITIS (Infections and infestations) | 1
HYPOKALEMIA (Vascular disorders) | 1
LEFT BUTTOCK ABSCESS (Infections and infestations) | 1
LACERATION OF SCALP (Injury, poisoning and procedural complications) | 1
RIGHT BREAST PAIN (Musculoskeletal and connective tissue disorders) | 1
HIP PAIN, RIGHT (Injury, poisoning and procedural complications) | 1
RIGHT CARPOMETACARPAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
OSTEOARTHRITIS LEFT KNEE (Musculoskeletal and connective tissue disorders) | 2
BILATERAL EYE CATARACT (Eye disorders) | 1
PAINFUL TOAL KNEE ARTHROPLASTY (RIGHT KNEE) (Musculoskeletal and connective tissue disorders) | 1
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 3
CARDIAC ARRHYTHMIA (Cardiac disorders) | 2
LEFT LATERAL EPICONDYLITIS (Musculoskeletal and connective tissue disorders) | 1
TINEA CORPORIS (Ear and labyrinth disorders) | 1
ILEITIS (Gastrointestinal disorders) | 1
PATELLAR TENDINITIS, RIGHT KNEE (Musculoskeletal and connective tissue disorders) | 1
INGUINAL HERNIA (Musculoskeletal and connective tissue disorders) | 1
EPIGASTRIC/CHEST PAIN (Gastrointestinal disorders) | 1
NASAL CONGESTION, COUGH (Respiratory, thoracic and mediastinal disorders) | 1
LEFT HIP PAIN (Injury, poisoning and procedural complications) | 7
INFLUENZA (Infections and infestations) | 2
ABDOMINAL PAIN, NAUSEA, DIARRHEA (Gastrointestinal disorders) | 1
ACUTE SUPPURATIVE OTITIS MEDIA OF RIGHT EAR WITHOUT SPONTANEOUS RUPTURE OF TYMPANIC MEMBRANE (Ear and labyrinth disorders) | 1
RIGHT FOOT EXTENSOR TENDONITIS (Injury, poisoning and procedural complications) | 1
RIGHT GLUTEAL PAIN (Musculoskeletal and connective tissue disorders) | 1
GERD WITHOUT ESOPHAGITIS (Gastrointestinal disorders) | 1
THROMBOSED HEMORRHOID (Gastrointestinal disorders) | 1
THROAT DISCOMFORT (Gastrointestinal disorders) | 1
PATIENT DIAGNOSED WITH CANCER, AGGRESSIVE. (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LEFT EYE PAIN, CORNEAL EROSION (Eye disorders) | 1
LAGOPHTHALMOS OF EYELIDS OF BOTH EYES (Eye disorders) | 1
SINUSITIS (Infections and infestations) | 1
ABRASION OF RIGHT CORNEA (Eye disorders) | 1
LUMBAR RADICULOPATHY, LOW BACK PAIN (Nervous system disorders) | 1
THORACIC RADICULOPATHY (Nervous system disorders) | 1
CALCULUS OF GALLBLADDER WITH ACUTE CHOLECYSTITIS (Blood and lymphatic system disorders) | 1
LEFT-SIDED NUMBNESS AND WEAKNESS (Injury, poisoning and procedural complications) | 1
HIGH STOMACH ACID (Gastrointestinal disorders) | 1
TRAVELER'S DIARRHEA (Gastrointestinal disorders) | 1
HEMORRHOIDS, EXTERNAL, THROMBOSED (Gastrointestinal disorders) | 1
CYST IN CERVICAL, OVARY, UTERUS (Injury, poisoning and procedural complications) | 1
ACUTE CHOLECYSTITIS (Hepatobiliary disorders) | 1
PELVIC AND LEFT HUMERUS FRACTURES DUE TO FALL (Injury, poisoning and procedural complications) | 1
STREPTOCOCOCCUS B (Infections and infestations) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 2
NAUSEA (Gastrointestinal disorders) | 1
UPPER GASTROINTESTINAL BLEEDING (Gastrointestinal disorders) | 1
LEFT HIP OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2
RIGHT GREAT TOE PAIN (HALLUX RIGIDUS) (Musculoskeletal and connective tissue disorders) | 1
RIGHT GREATER TROCHANTERIC PAIN SYNDROME (Injury, poisoning and procedural complications) | 1
SEIZURE, ENCEPHALOPATHY (Nervous system disorders) | 2
PELVIC PAIN (General disorders) | 2
ACUTE NONPERFORATED APPENDICITIS (Gastrointestinal disorders) | 1
TRAUMATIC ARTHRITIS OF RIGHT ANKLE (Musculoskeletal and connective tissue disorders) | 1
GASTRITIS WITH NAUSEA AND VOMITING (Gastrointestinal disorders) | 1
BILIARY COLIC (Hepatobiliary disorders) | 1
PERICOLONIC ABSCESS S/P APPENDECTOMY (Gastrointestinal disorders) | 1
GASTRITIS (Gastrointestinal disorders) | 1
VAGINAL ATROPHY (Reproductive system and breast disorders) | 1
HERNIA (Gastrointestinal disorders) | 1
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1
CLOSED FRACTURE OF DISTAL END OF RIGHT FIBULA (Musculoskeletal and connective tissue disorders) | 1
ACUTE CYSTITIS WITH HEMATURIA AND DYSURIA (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 1
HYPOTHYROIDISM (Endocrine disorders) | 1
ELEVATED BLOOD GLUCOSE LEVELS (Metabolism and nutrition disorders) | 1
PERSISTENT SEVERE HEADACHES (Nervous system disorders) | 1
NON-RECURRENT ACUTE SEROUS OTITIS MEDIA OF BOTH EARS (Ear and labyrinth disorders) | 1
VIRAL CONJUNCTIVITIS (Infections and infestations) | 1
ONYCHOMYCOSIS, RIGHT TOENAIL (Infections and infestations) | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2
DEHYDRATION (General disorders) | 1
VESTIBULAR MIGRAINES (Nervous system disorders) | 1
LEFT KNEE PAIN (Musculoskeletal and connective tissue disorders) | 8
SEVERE DEGENERATIVE JOINT DISEASE, RIGHT HIP (Musculoskeletal and connective tissue disorders) | 1
MELANOMA, NOSE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LEFT HIP PAIN (Musculoskeletal and connective tissue disorders) | 7
RIGHT GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1
DENTAL PAIN (Musculoskeletal and connective tissue disorders) | 1
RIGHT HAND PAIN AND FOREARM PAIN (Musculoskeletal and connective tissue disorders) | 1
RIGHT HIP ARTHRITIS (Musculoskeletal and connective tissue disorders) | 2
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
PAIN IN RIGHT SHOULDER (Musculoskeletal and connective tissue disorders) | 1
PHARYNGITIS AND RHINORRHEA (Respiratory, thoracic and mediastinal disorders) | 1
PHARYNGITIS WITH COUGH (Respiratory, thoracic and mediastinal disorders) | 1
LOW BACK PAIN (Musculoskeletal and connective tissue disorders) | 5
LEFT SHOULDER IMPINGEMENT,ACROMIOCLAVICULAR JOINT ARTHROSIS,BICEPS TENDINITIS & ROTATOR CUFF FRAYING (Musculoskeletal and connective tissue disorders) | 1
BICEPS TENDINITIS, LEFT (Musculoskeletal and connective tissue disorders) | 1
PAIN IN RIGHT WRIST (Musculoskeletal and connective tissue disorders) | 1
DYSLIPIDEMIA (Vascular disorders) | 1
SYPHILIS (Reproductive system and breast disorders) | 1
LEFT HAND PAIN (Musculoskeletal and connective tissue disorders) | 1
RIGHT HIP ARTHROPLASTY (TOTAL) FOR AVN (AVASCULAR NECROSIS) (Musculoskeletal and connective tissue disorders) | 1
FLUID LEVEL BEHIND TYMPANIC MEMBRANE OF BOTH EARS (Ear and labyrinth disorders) | 1
PINCHING SENSATION IN RIGHT HIP WHEN LIFTING HEAVY OBJECTS (Injury, poisoning and procedural complications) | 1
HYPERBILIRUBINEMIA (Vascular disorders) | 1
BILATERAL KNEE PAIN (Musculoskeletal and connective tissue disorders) | 2
ACUTE INTRACTABLE HEADACHE (Nervous system disorders) | 1
ALLERGIES (Vascular disorders) | 1
BAKER'S CYST BEHIND RIGHT KNEE AND SWELLING OF RIGHT KNEE (Musculoskeletal and connective tissue disorders) | 1
MIDLINE CYSTOCELE, PAIN IN FEMALE GENITALIA ON INTERCOURSE (Reproductive system and breast disorders) | 1
TRIGGER FINGER, LEFT HAND MIDDLE FINGER (Musculoskeletal and connective tissue disorders) | 1
DEGENERATIVE ARTHRITIS, RIGHT KNEE (Musculoskeletal and connective tissue disorders) | 1
TENDINITIS, RIGHT HIP (Musculoskeletal and connective tissue disorders) | 1
INSOMNIA (Nervous system disorders) | 1
BILATERAL FOOT PAIN (Musculoskeletal and connective tissue disorders) | 1
CLOSED FRACTURE OF MULTIPLE RIBS, LEFT SIDE (Musculoskeletal and connective tissue disorders) | 1
SHINGLES (Infections and infestations) | 1
RIGHT HIP DISLOCATION & THUMB CONTUSION W/O NAIL DAMAGE, CLOSED FRACTURE OF LEFT-SIDE MULTIPLE RIBS (Musculoskeletal and connective tissue disorders) | 1
RIGHT HIP FLEXOR TENDINITIS (Musculoskeletal and connective tissue disorders) | 1
OSTEOARTHRITIS, RIGHT KNEE (Musculoskeletal and connective tissue disorders) | 1
LEFT LOWER MEDIAL BREAST PAIN AND LUMP (Reproductive system and breast disorders) | 1
MUSCLE SPASMS (Injury, poisoning and procedural complications) | 3
HYPOVITAMINOSIS D (Vascular disorders) | 1
LIPOMA ON RIGHT LOWER EXTREMITY BELOW KNEE (Skin and subcutaneous tissue disorders) | 1
RIGHT HIP NOISE (Injury, poisoning and procedural complications) | 2
DEGENERATIVE ARTHRITIS, RIGHT HIP (Musculoskeletal and connective tissue disorders) | 1
LEFT GREATER TROCHANTERIC BURSITIS (Injury, poisoning and procedural complications) | 1
RIGHT HIP NOISE ASSOCIATED WITH NO PAIN (Injury, poisoning and procedural complications) | 1
HERPES ZOSTER WITHOUT COMPLICATION (Skin and subcutaneous tissue disorders) | 1
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1
POLYCYTHEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
POSITIVE COVID19 (Infections and infestations) | 1
LUMBAR SPONDYLOSIS, DEGENERATIVE DISC DISEASE, RADICULOPATHY (Nervous system disorders) | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 1
HALLUX RIGIDUS, RIGHT FOOT (Musculoskeletal and connective tissue disorders) | 1
LEFT HIP CLICKING AND SQUEAKING WITHOUT PAIN (Injury, poisoning and procedural complications) | 1
NECK PAIN, LOW BACK PAIN (Musculoskeletal and connective tissue disorders) | 1
LEFT AND RIGHT KNEE PAIN (Musculoskeletal and connective tissue disorders) | 1
BILATERAL TARSOMETATARSAL ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
WOUND INFECTION, RIGHT LOWER LEG (Infections and infestations) | 1
LUMBAR STENOSIS (Nervous system disorders) | 1
OSTEOARTHRITIS, RIGHT HIP (Musculoskeletal and connective tissue disorders) | 2
SACROILIITIS, UNKNOWN SIDE (Injury, poisoning and procedural complications) | 1
ARTHRITIS, RIGHT HIP (Musculoskeletal and connective tissue disorders) | 1
LEFT ANKLE PAIN (Musculoskeletal and connective tissue disorders) | 2
PAIN IN RIGHT KNEE, RIGHT KNEE OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
RIGHT HIP OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
LUNG CANCER, LEFT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LEFT HEEL PAIN (Musculoskeletal and connective tissue disorders) | 1
TROCHANTERIC BURSITIS, BILATERAL (Injury, poisoning and procedural complications) | 1
RIGHT HIP PAIN (Musculoskeletal and connective tissue disorders) | 8
HEADACHES (Nervous system disorders) | 1
RIGHT HIP PAIN (Injury, poisoning and procedural complications) | 8
SEVERE ACUTE RESPIRATORY SYNDROME CORONAVIRUS 2 (Infections and infestations) | 1
SOLITARY BRAIN METASTASIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LEFT HIP SORENESS AND POPPING (Injury, poisoning and procedural complications) | 1
BILATERAL PTOSIS OF UPPER EYELIDS (Eye disorders) | 1
FREQUENT NIGHT URINATION (Renal and urinary disorders) | 1
LEFT HIP POSTOPERATIVE PAIN (Injury, poisoning and procedural complications) | 1
MIXED HYPERLIPIDEMIA (Vascular disorders) | 1
SLEEP APNEA (Nervous system disorders) | 1
LEFT LOWER BACK PAIN (Musculoskeletal and connective tissue disorders) | 1
CERVICAL RADICULOPATHY WITH NUMBNESS AND TINGLING OF LEFT HAND (Nervous system disorders) | 1
LEFT KNEE OSTEOARTHRITIS, LEFT KNEE PAIN (Musculoskeletal and connective tissue disorders) | 1
ELEVATED GLUCOSE (Vascular disorders) | 1
LOW HIGH DENSITY LIPOPROTEIN LEVEL (Vascular disorders) | 1
PAIN IN LEFT SHOULDER (Musculoskeletal and connective tissue disorders) | 1
RIGHT HIP PAIN AND DISCOMFORT (Musculoskeletal and connective tissue disorders) | 1
RIGHT HIP PAIN POST-OP LAMINECTOMY (Injury, poisoning and procedural complications) | 1
INGROWN TOENAIL ON LEFT BIG TOE (Skin and subcutaneous tissue disorders) | 1
RIGHT HIP PAIN SECONDARY TO OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
POSTERIOR NECK LIPOMA (Skin and subcutaneous tissue disorders) | 1
RIGHT HIP SORENESS AND NOISE (Injury, poisoning and procedural complications) | 1
SEVERE ACUTE SYNDROME CORONAVIRUS 2 (Infections and infestations) | 1
ALLERGIC REACTION TO ORAL RIVAROXABAN (Vascular disorders) | 1
RIGHT HIP TROCHANTERIC BURSITIS (Injury, poisoning and procedural complications) | 1
GANGLION CYST OF TENDON SHEATH OF RIGHT HAND (Musculoskeletal and connective tissue disorders) | 1
RIGHT ILIOPSOAS TENDINITIS (Musculoskeletal and connective tissue disorders) | 1
RIGHT INTRAOPERATIVE CALCAR FRACTURE (Musculoskeletal and connective tissue disorders) | 1
HYPERLIPIDEMIA (Vascular disorders) | 2
LEFT HIP PAIN SECONDARY TO OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 3
RIGHT IT BAND TENDINITIS, GREATER TROCHANTERIC BURSITIS (Injury, poisoning and procedural complications) | 1
LEFT NECK PAIN AND SWELLING OF PORT CATHETER (Injury, poisoning and procedural complications) | 1
CHEST PAIN (General disorders) | 1
TROCHANTERIC BURSITIS OF RIGHT HIP (Injury, poisoning and procedural complications) | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 2
LEFT HIP PAIN / PRIMARY OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
LUPUS (EARLY STAGE DIAGNOSIS) (Vascular disorders) | 1
LEFT ELBOW PAIN (Musculoskeletal and connective tissue disorders) | 1
ACUTE LOW BACK PAIN DUE TO A FALL (Injury, poisoning and procedural complications) | 1
RIGHT IT BAND TIGHTNESS (Musculoskeletal and connective tissue disorders) | 1
FAILED TOTAL HIP JOINT (RIGHT SIDE) (Product Issues) | 1
RIGHT KNEE ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
RIGHT KNEE PAIN (Injury, poisoning and procedural complications) | 4
POST-OP FEVERS (General disorders) | 1
LEFT HEEL AND FOOT PAIN AND SWELLING (Musculoskeletal and connective tissue disorders) | 1
ANKLE PAIN, LEFT (Musculoskeletal and connective tissue disorders) | 1
RIGHT KNEE PAIN (Musculoskeletal and connective tissue disorders) | 4
SPINAL STENOSIS (Nervous system disorders) | 1
ILIOPSOAS TENDINITIS OF THE LEFT HIP (Musculoskeletal and connective tissue disorders) | 1
GREATER TROCHANTERIC BURSITIS, RIGHT HIP (Injury, poisoning and procedural complications) | 1
OSTEOARTHRITIS, LEFT KNEE (Musculoskeletal and connective tissue disorders) | 2
POST-OPERATIVE SQUEAKING, LEFT HIP (Injury, poisoning and procedural complications) | 1
PRIMARY OPEN-ANGLE GLAUCOMA, BILATERAL (Eye disorders) | 1
RIGHT KNEE PAIN - UNILATERAL PRIMARY KNEE OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
RIGHT LOWER EXTREMITY PAIN AND SWELLING (Musculoskeletal and connective tissue disorders) | 1
CALCAR FRATURE INTRAOPERATIVELY (Injury, poisoning and procedural complications) | 1
SUPRAPATELLAR BURSITIS OF LEFT KNEE (Injury, poisoning and procedural complications) | 1
RIGHT LUNG LOWER LOBE PULMONARY NODULE (Respiratory, thoracic and mediastinal disorders) | 1
OSTEOARTHRITIS OF MCP JOINT, RIGHT THUMB (Musculoskeletal and connective tissue disorders) | 1
LEFT KNEE PAIN SECONDARY TO FALL (Injury, poisoning and procedural complications) | 1
RIGHT OLECRANON BURSITIS (Injury, poisoning and procedural complications) | 1
WORSENING RIGHT SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 1
GLENOHUMERAL JOINT OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
PAIN AT INCISION SITE (Injury, poisoning and procedural complications) | 1
RIGHT PSOAS TENDINITIS (Musculoskeletal and connective tissue disorders) | 1
KNEE OSTEOARTHRITIS, BILATERAL (Musculoskeletal and connective tissue disorders) | 1
RIGHT RING TRIGGER FINGER, LEFT WRIST DE QUERVAIN'S (Musculoskeletal and connective tissue disorders) | 1
LEFT ANKLE FRACTURE (DISTAL FIBULA) (Musculoskeletal and connective tissue disorders) | 1
WORSENING LEFT KNEE PAIN SECONDARY TO OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2
MILD TRAUMA TO OPERATIVE HIP. PATIENT BUMPED INTO METAL POLE. (Injury, poisoning and procedural complications) | 1
GOUT. LEFT ANKLE (Musculoskeletal and connective tissue disorders) | 1
TORN ROTATOR CUFF (Musculoskeletal and connective tissue disorders) | 1
FALL (Injury, poisoning and procedural complications) | 2
RIGHT SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 3
TYPHOID FEVER - PNEUMONIA (Infections and infestations) | 1
LEFT TROCHANTERIC BURSITIS (Injury, poisoning and procedural complications) | 1
SEVERE RIGHT HIP OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2
ILIOPSOAS TENDINITIS (Musculoskeletal and connective tissue disorders) | 1
LEFT HIP OSTEOARTHRITIS - WORSENING PAIN (Musculoskeletal and connective tissue disorders) | 1
PRIMARY OSTEOARTHRITIS LEFT HIP (Musculoskeletal and connective tissue disorders) | 1
HIP OSTEOARTHRITIS (LEFT HIP) (Musculoskeletal and connective tissue disorders) | 1
LEFT KNEE OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
SHINGLES (VARICELLA ZOSTER) (Skin and subcutaneous tissue disorders) | 1
BRAIN TUMOR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LUMBAR BACK PAIN (Musculoskeletal and connective tissue disorders) | 1
MINOR FALL (Injury, poisoning and procedural complications) | 1
PROXIMAL BICEPS TENDINOPATHY RIGHT SHOULDER (Musculoskeletal and connective tissue disorders) | 1
TRAUMATIC INJURY OF HEAD (Injury, poisoning and procedural complications) | 1
NEUROPLASTY RIGHT CARPAL TUNNEL RELEASE DUE TO ARTHRITIS OF CARPOMETACARPAL (Musculoskeletal and connective tissue disorders) | 1
FOLLOW-UP BILATERAL HIP DISCOMFORT (Musculoskeletal and connective tissue disorders) | 1
AVASCULAR NECROSIS OF BONE OF LEFT HIP (Musculoskeletal and connective tissue disorders) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1
RIGHT SHOULDER ROTATOR CUFF ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1
RIGHT THIGH NUMBNESS (Nervous system disorders) | 1
LEFT TOTAL KNEE REPLACEMENT DUE TO POST-TRAUMATIC ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
OSTEOARTHRITIS IN RIGHT HIP (Musculoskeletal and connective tissue disorders) | 2
WORSENING RIGHT LEG PAIN (Musculoskeletal and connective tissue disorders) | 1
BILATERAL LOW BACK PAIN WITHOUT SCIATICA (Musculoskeletal and connective tissue disorders) | 1
LUMBAR DEGENERATIVE DISC DISEASE (Nervous system disorders) | 1
SWELLING LEFT IN HIP (Musculoskeletal and connective tissue disorders) | 1
RIGHT THIGH PAIN (Musculoskeletal and connective tissue disorders) | 1
INCREASED LEFT HIP PAIN (Musculoskeletal and connective tissue disorders) | 1
PAIN FOR RIGHT TOTAL HIP ARTHROPLASTY (Musculoskeletal and connective tissue disorders) | 1
INCREASED/WORSENING RIGHT HIP PAIN OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
FEVER (General disorders) | 1
STAGE 2 KIDNEY DISEASE (Renal and urinary disorders) | 1
FREQUENT EPISTAXIS (Gastrointestinal disorders) | 1
LEFT HIP BURSITIS (Musculoskeletal and connective tissue disorders) | 1
LEFT BUNION WITH ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
LEFT BASILAR JOINT ARTHRITIS OF THE THUMB (Musculoskeletal and connective tissue disorders) | 1
BILATERAL SHOULDER ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
CERVICAL MYELORADICULOPATHY (Musculoskeletal and connective tissue disorders) | 1
END STAGE RIGHT SHOULDER ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
PSOAS TENDINITIS, RIGHT (Musculoskeletal and connective tissue disorders) | 1
WORSENING LEFT KNEE OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
FALL INVOLVING RIGHT HIP (Injury, poisoning and procedural complications) | 1
PURE HYPERCHOLESTEROLEMIA (Vascular disorders) | 1
WORSENING LEFT HIP OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
BURSITIS IN RIGHT HIP (Injury, poisoning and procedural complications) | 1
CRAMPS, MUSCLE SPASM (Musculoskeletal and connective tissue disorders) | 1
WORSENING RIGHT HIP OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
FACIAL LESION (Skin and subcutaneous tissue disorders) | 1
ALLERGIC REACTION (RASH) ON TRUNK OF BODY. (Skin and subcutaneous tissue disorders) | 1
ADVERSE DRUG REACTION TO BACTRIM (Injury, poisoning and procedural complications) | 1
BILATERAL HIP PAIN DUE TO ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1
MUSCLE SPASM AND ILIOPSOAS TENDINITIS (Musculoskeletal and connective tissue disorders) | 1
WORSENING NEPHROTIC SYNDROME (Renal and urinary disorders) | 1
RIGHT TOTAL KNEE REPLACEMENT (Musculoskeletal and connective tissue disorders) | 1
WORSENING CONGENITAL DYSPLASIA LEFT HIP (Congenital, familial and genetic disorders) | 1
DEATH DUE TO DRUG OVERDOSE (Injury, poisoning and procedural complications) | 1
FRACTURED LEFT ANKLE (Musculoskeletal and connective tissue disorders) | 1

LIMITATIONS AND CAVEATS:
The impact of the COVID-19 pandemic on participant retention, out of window follow-up visits, and data acquisition due to participants being unable or not willing to undergo study assessments at follow-up visits. Primary outcome analyses were not impacted by COVID-19. Data missing for secondary outcome analyses was low and risks were mitigated by appropriate alternative data collection methods.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period up to 90 days but less than or equal to 180 days from the time submitted to the sponsor for review. Sponsor may delay publication up to 180 days to permit the filing of appropriate patent applications if the sponsor believes any publication contains any information relating to patentable items and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2023-12-14): https://cdn.clinicaltrials.gov/large-docs/34/NCT03056534/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-19): https://cdn.clinicaltrials.gov/large-docs/34/NCT03056534/SAP_001.pdf